CLINICAL TRIAL: NCT04438278
Title: Neutropenic Enterocolitis in Critically Ill Hematological Patients: Taxonomic and Functional Analysis of Gut Microbiota
Brief Title: Profile Fecal Analysis of Neutropenic Enterocolitis
Acronym: PROFANE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190826
Record Dates: First submitted 2020-05-26; First posted 2020-06-18 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Neutropenic Enterocolitis
MeSH Terms: conditions — Enterocolitis, Neutropenic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective, single-center, cohort study to allow collecting observations of patients receiving induction chemotherapy for primary Acute Myeloid Leukemia (AML), collecting biological samples(including fecal samples for microbiota analyses, and metagenomic profiling in blood samples) and clinical outcomes (notably the occurrence of neutropenic enterocolitis), with a nested case-control analysis comparing patients with or without neutropenic enterocolitis

ELIGIBILITY:
Inclusion Criteria:

* patient>= 18 years old;
* cytological diagnosis of de novo Acute Myeloid Leukemia (AML) (>20% myeloid blasts);
* eligible for intensive chemotherapy (no severe co-morbidity);
* not having received any prior chemotherapy;
* affiliation to the national social security system.

Exclusion Criteria:

* acute promyelocytic leukemia (AML 3);
* inability to understand the nature of investigations or to give informed non-opposition;
* person subject to a legal protection measure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients receiving induction chemotherapy for primary Acute Myeloid Leukemia (AML)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2022-07-08 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Shannon index of α-diversity | At day 1, before chemotherapy initiation
  Shannon index of α-diversity assessed by shotgun metagenomic analysis of the stool

SECONDARY OUTCOMES:
Fecal microbiota's profile | At day 14
  Taxonomic identification in shotgun metagenomic
Intensive Care Unit (ICU) - mortality | 60 days
  Death while hospitalized in the intensive care unit
Hospital - mortality | 60 days
  Death while hospitalized
1-year mortality | 1 year
  Death within 1 year of inclusion
Occurrence of any local neutropenic enterocolitis complications | 60 days
  Local neutropenic enterocolitis complications defined as perforation or digestive hemorrhage or abscess
Occurrence of microbiologically documented infections in patients with severe neutropenic enterocolitis | 60 days
  Microbiologically documented infections defined as pneumonia, invasive device infections, urinary tract infections, digestive or neuro-meningitis infections
Occurrence of malnutrition in patients with severe neutropenic enterocolitis | 60 days
  Malnutrition defined by the European Society of Clinical nutrition and Metabolism
Biodiversity in microbiota | Day 1, day 14, day 28, day 42
  Analysis of alpha and beta-diversity in fecal samples from day 0 to day 60
Whole-blood metatranscriptomic profile evolution | Day 1, day 14, day 28, day 42
  Identification of clusters of gene expression

CONTACTS AND LOCATIONS:
Locations (1):
- AP-HP Hôpital Saint Louis, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kapandji N, Salmona M, Lemoine A, Ulmann G, Calderaro J, Roche B, Kapel N, Biard L, Lengline E, Goff JL, Rodriguez C, Thomas M, Zafrani L. Unravelling neutropenic enterocolitis: insights from gut microbiota, and intestinal barrier analyses. Exp Hematol Oncol. 2025 May 16;14(1):74. doi: 10.1186/s40164-025-00661-4. PMID 40380332